CLINICAL TRIAL: NCT03387670
Title: A Phase 3 Randomised, Double Blind, Clinical Trial Investigating the Effectiveness of Repurposed Simvastatin Compared to Placebo, in Secondary Progressive Multiple Sclerosis, in Slowing the Progression of Disability
Brief Title: Multiple Sclerosis-Simvastatin Trial 2
Acronym: MS-STAT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University of Edinburgh (Other); Queen Mary University of London (Other); London School of Hygiene and Tropical Medicine (Other); University of Leeds (Other); The Leeds Teaching Hospitals NHS Trust (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17/0158; 2017-003328-56 (EudraCT Number)
Record Dates: First submitted 2017-11-28; First posted 2018-01-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Secondary Progressive Multiple Sclerosis (SPMS)
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — * One (1 = 40mg) simvastatin tablet once daily at night for 1 month
  * Two (2 = 80mg) simvastatin tablets once daily at night, for the next 35 to 53 months
  Arms: Simvastatin
Drug: Placebo — * One (1) placebo tablet once daily at night for 1 month
  * Two (2) placebo tablets once daily at night, for the next 35 to 53 months
  Arms: Placebo

SUMMARY:
Multiple Sclerosis (MS) is a progressive neurological disorder of the brain and spinal cord. It affects approximately 120,000 people in the United Kingdom and 2.5 million people globally. Most people with MS experience two stages of the disease:

Early MS - Relapsing-Remitting MS (RRMS), which is partially reversible, and Late MS - Secondary Progressive MS (SPMS), which affects the majority of patients, usually after 10 to 15 years after diagnosis.

SPMS results from progressive neuronal degeneration that causes accumulating and irreversible disability affecting walking, balance, manual function, vision, cognition, pain control, bladder and bowel function. The pathological process driving the accrual of disability in SPMS is not known at present.

Immunomodulatory anti-inflammatory disease modifying therapies (DMTs) are increasingly effective in reducing relapse frequency in RRMS, however, they have been unsuccessful in slowing disease progression in SPMS. This is the overwhelming conclusion from an analysis of 18 phase 3 trials (n=8500), of which 70% of the population had SPMS, all performed in the last 25 years.

In an earlier study (Multiple Sclerosis-Simvastatin 1; MS-STAT1), 140 people with SPMS were randomly assigned to receive either placebo or simvastatin for a period of two years. The investigators found that the rate of brain atrophy (loss of neurons - 'brain shrinkage'), as measured by magnetic resonance imaging (MRI), was reduced in patients receiving simvastatin compared to those taking placebo.

Several other long term studies have also reported that there might be a relationship between the rate of brain atrophy and the degree of impairment. The study is designed to test the effectiveness of repurposed simvastatin (80mg) in a phase 3 double blind, randomised, placebo controlled trial (1:1) in patients with secondary progressive MS (SPMS), to determine if the rate of disability progression can be slowed over a 3 to 4.5 year period.

The results generated from this trial may help to improve the treatment options of people with MS. In addition, taking part in this trial will mean regular review by an experienced neurologist regardless of the drug that patients are randomly allocated to receive.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of multiple sclerosis (MS) that have entered the secondary progressive stage. Steady progression rather than relapse must be the major cause of increasing disability in the preceding 2 years. Progression can be evident from either an increase of at least 1 point if EDSS score <6, or an increase of 0.5 point if EDSS score ≥6, or clinical documentation of increasing disability;
2. EDSS 4.0 - 6.5 (inclusive);
3. Aged 25 to 65 years old;
4. Patients must be able and willing to comply with the terms of this protocol;
5. Written informed consent provided.

Exclusion Criteria:

1. Relapse within 3 months of baseline visit. Patients will be eligible where 3 months from the final day of the relapse, has elapsed by the date of the baseline visit;
2. Patients that have been treated with steroids (intravenous and/or oral) due to MS relapse/progression within 3 months from the final day of relapse to the baseline visit. These patients may undergo a further screening visit once the 3 month window has expired and may be included if no steroid treatment has been administered in the intervening period; (Note: Patients on steroids for another medical condition may be included in the trial provided the steroid prescription is not for MS relapse/progression)
3. Significant organ co-morbidity e.g. cardiac failure, renal failure, malignancy;
4. Screening levels of alanine aminotransferase (ALT) / aspartate aminotransferase (AST) or creatine kinase (CK) ≥3 x upper limit of normal (ULN);
5. Current use of a statin; or any use within the last 6 months;
6. Medications that interact unfavourably with simvastatin as outlined in the current summary of product characteristics (SmPC); including but not limited to CYP3A4 inhibitors (e.g. itraconazole, ketoconazole, posaconazole, voriconazole, fluconazole, HIV protease inhibitors (e.g. nelfinavir), boceprevir, erythromycin, clrithromycin, telithromycin, telaprevir, nefazodone, fibrates (including fenofibrates), nicotinic acid (or products containing niacin), azole anti-fungal preparations, macrolide antibiotics, protease inhibitors, verapamil, amiodarone, amlodipine, gemfibrozil, ciclosporin, danazol, diltiazem, rifampicin, fusidic acid, elbasvir, grazoprevir,ticagrelor, daptomycin, grapefruit juice or alcohol abuse;
7. Primary progressive MS;
8. Diabetes mellitus type 1;
9. Uncontrolled hypothyroidism;
10. Female participants that are pregnant or breast feeding. Women of child bearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period, and up to 4 weeks after the last dose of study drug;
11. Use of immunosuppressants (e.g. azathioprine, methotrexate, ciclosporine) or disease modifying treatments (avonex, rebif, betaferon, glatiramer) within the previous 6 months;
12. Use of mitoxantrone, natalizumab, alemtuzumab, daclizumab or other monoclonal antibody treatment, if treated within the last 12 months;
13. Use of fingolimod, dimethyl fumarate, teriflunomide, cladribine within the last 12 months;
14. Use of other experimental disease modifying treatment within the last 6 months;
15. Commencement of fampridine ≤6 months from day of randomisation;
16. Concurrent participation in another clinical trial of an investigational medicinal product or medical device;
17. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Time to confirmed disability progression between simvastatin and placebo arm based on change in EDSS scores compared to baseline. | 6 monthly - baseline, month 6, 12, 18, 24, 30, 36, 42, 48, 54
  The initial disability progression event is finalised as positive if disability is sustained and confirmed ≥6* months later. Progression of disability defined as an increase of at least 1 point if EDSS baseline score <6, or an increase of 0.5 point if baseline EDSS score is ≥6.

SECONDARY OUTCOMES:
Response rate on the patient reported outcome form Multiple Sclerosis Walking Scale-12 version 2 (MSWS-12v2) | Annually - baseline, month 12, 24 and 36
  MSWS-12v2 is a12 item patient report measure on the impact of MS on the individual's walking ability over the previous 2 weeks. Each item will be summed to generate a total score and transformed to a scale with a range of 0 to 100 with high scores indicating greater impact on walking.
Response rate on the patient reported outcome form Multiple Sclerosis Impact Scale-29 version 2 (MSIS-29v2) | Annually - baseline, month 12, 24 and 36
  MS Impact Scale-29 version 2 (MSIS-29v2) - A psychometrically validated patient-reported outcome measure increasingly used for measuring the impact of MS on people's lives. The 29-item scale assesses the impact of MS on people's health related quality of life in terms of their physical and psychological well-being over the previous 2 weeks.
Cost effectiveness of intervention | 6 monthly - baseline, month 6, 12, 18, 24, 30, 36
  To estimate the incremental cost and cost-effectiveness of simvastatin versus standard care for the trial period and for the lifetime horizon using the Client Client Services Receipt Inventory Form.
Evaluating change in degree of disability based on the modified Rankin scale (mRS) | Annually - baseline, month 12, 24 and 36
  mRS is used to evaluate the degree of disability in daily activities of those with neurological disability.
Change in visual function based on the Sloan Low Contrast Visual Acuity (SLCVA) | Annually - baseline, month 12, 24 and 36
  Sloan chart testing is a reliable, quantitative, and clinically practical measure of visual function that will be administered by trained assessors. The chart consists of rows of grey letters on a white background. Letters are displayed in decreasing order from the top of the chart to the bottom. Testing will be conducted at three different contrast levels (100%, 2.5% and 1.25%). The chart will be scored based on the number of letters correctly identified out of 60.
Difference in patient reported quality of life based on the EuroQoL Health Related Quality of Life - 5 Dimensions - 5 Levels (EQ-5D 5L) scores | 6 monthly - baseline, month 6, 12, 18, 24, 30, 36
  EQ-5D 5L is a 5 item questionnaire (assessing - mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and visual analogue scale (VAS) enables calculation of quality adjusted life years (QALY) to enable health economic analyses to be performed. Each dimension assessed has 5 response scales to select from: no problems, slight problems, moderate problems, severe problems, and extreme problems
Change in a modified Multiple Sclerosis Functional Composite scores | Annually - baseline, month 12, 24 and 36
  A Modified Multiple Sclerosis Functional Composite (MSFC) score comprised of 3 components (T25FW, 9HPT, SDMT). The Symbol digit modalities test (SDMT) will replace the Paced Auditory Serial Addition Test (PASAT), one of the three components in the Standard MSFC.
Change in cognitive performance as measured by Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) | Baseline and month 36
  BICAMS is a composite cognitive assessment tool comprising of the three components : Symbol Digit Modalities Test (SDMT) , California Verbal Learning Test-II (CVLT-II) and Brief visuospatial memory test- Revised (BVMT-R)
Change in cognitive impairment based on Symbol Digit Modalities Test (SDMT) scores | Annually - baseline, month 12, 24 and 36
  SDMT is a brief measure of cognitive processing speed. It measures information processing speed for visually presented stimuli, but is self-paced, with at least equal reliability and sensitivity to the presence of worsening cognitive impairment.
Change in fatigue as measured by the Chalder Fatigue Scale | Annually - baseline, month 12, 24 and 36
  A questionnaire measuring the severity of physical and mental fatigue. The total score range is minimum of 0 and maximum of 33.
  For the subscales, physical fatigue score has a minimum of 0 and maximum of 21. The Mental fatigue score has a minimum of 0 and maximum of 12.
Change in rates of service utilisation as measured by the Client Service Receipt Inventory (CSRI) questionnaire | 6 monthly - baseline, month 6, 12, 18, 24, 30, 36
  The CSRI is a questionnaire that collects information on service utilisation, income, accommodation and other cost-related variables. Its primary purpose is to allow resource use patterns in each of the two arms to be described, and support costs to be estimated for health economics purposes.
Change in time taken to complete 25-Foot Timed Walk (T25FW) | 6 monthly - baseline, month 6, 12, 18, 24, 30, 36, 42, 48, 54
  T25-FW is a quantitative mobility and leg function performance test based on a timed 25-foot walk
Difference in the number and severity of multiple sclerosis related relapse events between treatment groups | 6 monthly - baseline, month 6, 12, 18, 24, 30, 36, 42, 48, 54
  A relapse will be defined as new or worsening neurological symptom(s) in the absence of fever, lasting for more than 24 hours, and have been preceded by a period of clinical stability of at least 30 days, with no other explanation than MS.
Evaluating the time to disability progression based on a secondary composite progression outcome measure | 6 monthly - baseline, month 6, 12, 18, 24, 30, 36, 42, 48, 54
  A secondary composite progression outcome measure defined as one or more of: ≥20% increase in time taken to complete the 25 Foot Walk (T25FW); or ≥20% increase in time to complete 9 Hole Peg Test (9HPT); or increase in EDSS (0.5 point increase if baseline ≥6 /1.0 point increase if baseline <6). The initial disability progression event will be finalised as positive if it is sustained and confirmed ≥6 months later*. The time to event analysis will be from randomisation until date of the initial disability progression (if subsequently confirmed)
Change in time taken to complete 9 hole peg test (9HPT) | 6 monthly - baseline, month 6, 12, 18, 24, 30, 36, 42, 48, 54
  The 9HPT is a brief, standardized, quantitative test of upper extremity function. Participants are instructed to pick up 9 pegs, one at a time, as quickly as possible and are required to insert them into 9 empty peg holes. Once all nine pegs have been inserted, the participant should immediately remove the pegs, one at a time. The total time taken to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The two trials for each hand are averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Chataway, Principal Investigator — University College, London
Locations (31):
- United Kingdom (31):
  - Belfast City Hospital, Belfast
  - St Luke s Hospital, Bradford
  - Royal Sussex County Hospital, Brighton
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - University Hospital of Wales, Cardiff
  - University Hospital Coventry and Warwickshire, Coventry
  - The Anne Rowling Regenerative Neurology Clinic, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - The Queen Elizabeth University Hospital, Glasgow
  - Hull Royal Infirmary, Hull
  - Leeds General Infirmary, Leeds
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Queen's Hospital, Barking, Havering and Redbridge University Hospitals, London
  - Queen Elizabeth Hospital, London
  - Charing Cross Hospital, London
  - University College London Hospital, London
  - Salford Royal Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich
  - Queen's Medical Centre, Nottingham
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Poole Hospital, Poole
  - Royal Preston Hospital, Preston
  - Royal Hallamshire Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - University Hospital of North Staffordshire, Stoke-on-Trent
  - Morriston & Neath Port Talbot Hospitals (Abertawe Bro Morgannwg University Local Health Board), Swansea
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chataway J, Williams T, Blackstone J, John N, Braisher M, De Angelis F, Bianchi A, Calvi A, Doshi A, Apap Mangion S, Wade C, Bordea E, Merry R, Barton G, Lyle D, Jarman E, Mahad D, Shehu A, Arun T, McDonnell G, Geraldes R, Craner M, Hillier C, Ganesalingam J, Fisniku L, Hobart J, Spilker C, Robertson NP, Kalra S, Pluchino S, Harikrishnan S, Mattoscio M, Harrower T, Young C, Lee M, Chhetri SK, Ahmed F, Rog D, Silber E, Gallagher P, Duddy M, Straukiene A, Nicholas R, Rice C, Tebbs S, Hawton A, Hunter R, Giovannoni G, Ciccarelli O, Beveridge J, Nixon S, Thompson AJ, Greenwood J, Pearson OR, Evangelou N, Sharrack B, Galea I, Gray E, Pavitt S, Chandran S, Ford HL, Frost C, Nicholas JM; MS-STAT2 Investigators. Effect of repurposed simvastatin on disability progression in secondary progressive multiple sclerosis (MS-STAT2): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2025 Oct 11;406(10512):1611-1624. doi: 10.1016/S0140-6736(25)01039-6. Epub 2025 Oct 1. PMID 41045938
- [Derived] Blackstone J, Williams T, Nicholas JM, Bordea E, De Angelis F, Bianchi A, Calvi A, Doshi A, John N, Apap Mangion S, Wade C, Merry R, Barton G, Lyle D, Jarman E, Mahad D, Shehu A, Arun T, McDonnell G, Geraldes R, Craner M, Hillier C, Ganesalingam J, Fisniku L, Hobart J, Spilker C, Robertson N, Kalra S, Pluchino S, Harikrishnan S, Mattoscio M, Harrower T, Young C, Lee M, Chhetri S, Ahmed F, Rog D, Silber E, Gallagher P, Duddy M, Straukiene A, Nicholas R, Rice C, Nixon SJ, Beveridge J, Hawton A, Tebbs S, Braisher M, Giovannoni G, Ciccarelli O, Greenwood J, Thompson AJ, Hunter R, Pavitt S, Pearson O, Evangelou N, Sharrack B, Galea I, Chandran S, Ford HL, Frost C, Chataway J. Evaluating the effectiveness of simvastatin in slowing the progression of disability in secondary progressive multiple sclerosis (MS-STAT2): protocol for a multicentre, randomised controlled, double-blind, phase 3 clinical trial in the UK. BMJ Open. 2024 Sep 16;14(9):e086414. doi: 10.1136/bmjopen-2024-086414. PMID 39284697
- [Derived] Williams T, John N, Calvi A, Bianchi A, De Angelis F, Doshi A, Wright S, Shatila M, Yiannakas MC, Chowdhury F, Stutters J, Ricciardi A, Prados F, MacManus D, Braisher M, Blackstone J, Ciccarelli O, Gandini Wheeler-Kingshott CAM, Barkhof F, Chataway J; UCL MS-STAT2 investigators. Cardiovascular risk factors in secondary progressive multiple sclerosis: A cross-sectional analysis from the MS-STAT2 randomized controlled trial. Eur J Neurol. 2023 Sep;30(9):2769-2780. doi: 10.1111/ene.15924. Epub 2023 Jun 23. PMID 37318885
- [Derived] Williams T, Tur C, Eshaghi A, Doshi A, Chan D, Binks S, Wellington H, Heslegrave A, Zetterberg H, Chataway J. Serum neurofilament light and MRI predictors of cognitive decline in patients with secondary progressive multiple sclerosis: Analysis from the MS-STAT randomised controlled trial. Mult Scler. 2022 Oct;28(12):1913-1926. doi: 10.1177/13524585221114441. Epub 2022 Aug 9. PMID 35946107
- [Derived] Williams T, Alexander S, Blackstone J, De Angelis F, John N, Doshi A, Beveridge J, Braisher M, Gray E, Chataway J; MS-SMART and MS-STAT2 Investigators. Optimising recruitment in clinical trials for progressive multiple sclerosis: observational analysis from the MS-SMART and MS-STAT2 randomised controlled trials. Trials. 2022 Aug 9;23(1):644. doi: 10.1186/s13063-022-06588-z. PMID 35945550
- [Derived] Williams TE, Holdsworth KP, Nicholas JM, Eshaghi A, Katsanouli T, Wellington H, Heslegrave A, Zetterberg H, Frost C, Chataway J. Assessing Neurofilaments as Biomarkers of Neuroprotection in Progressive Multiple Sclerosis: From the MS-STAT Randomized Controlled Trial. Neurol Neuroimmunol Neuroinflamm. 2022 Jan 14;9(2):e1130. doi: 10.1212/NXI.0000000000001130. Print 2022 Mar. PMID 35031587